CLINICAL TRIAL: NCT02551848
Title: Botulinum Toxin Type A for Injection of Bilateral Upper Extremity Tremor in Patients With Essential Tremor Using Kinematic Assessment
Brief Title: Kinematic-based BoNT-A Injections for Bilateral ET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Principal Investigator, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104584
Record Dates: First submitted 2015-09-11; First posted 2015-09-16 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Essential Tremor
Keywords: Movement disorders; Botulinum toxin type A; Kinematics
MeSH Terms: conditions — Essential Tremor; Movement Disorders | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Essential tremor treatment (Experimental): A serotype of botulinum toxin type A (BoNT-A) that has specificity for cleavage of SYNAPTOSOMAL-ASSOCIATED PROTEIN 25 (SNAP-25). BoNT-A's pharmacological action is to inhibit the release of acetylcholine from the neuromuscular junction.
  Participants will be treated by BoNT-A injections every 12 weeks over 72 weeks. BoNT-A parameters will be determined solely by biomechanical analysis of tremulous movements in both upper extremity BoNT-A dose will range from 50-300 U per arm
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A
  Other Names: IncobotulinumtoxinA; BoNT-A; Xeomin

SUMMARY:
The primary objective is to study the efficacy of botulinum toxin type A (Xeomin®) injected utilizing kinematically-based injection parameters for the treatment of upper extremity essential tremor (ET). Additional objectives are to study the benefit of kinematic assessment tools in determining injection parameters and to study the composition of tremor using kinematics.

ELIGIBILITY:
Inclusion Criteria:

* Consenting male and female participants
* Diagnosis of 'definite essential tremor' in accordance with the TRIG criteria including: ET individuals diagnosed with upper limb tremor in their motor dominant and non-dominant hands
* Stable ET medication management for the 3 month duration prior to their enrollment in the study
* Participants who are botulinum toxin naïve for tremor management
* Patients will be screened for pregnancy by the physician

Exclusion Criteria:

* History of stroke
* Muscle weakness or any related compartmental muscle syndrome
* Smoking
* History of ALS or Myasthenia Gravis
* Offending medications (Lithium, valproate, steroids, amiodarone, beta-adrenergic agonists (e.g. salbutamol)
* Persons prescribed zonisamide
* History of allergic or side effect reaction to botulinum toxin
* Contraindications per the Xeomin® drug monograph
* Women reporting that they are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Kinematic tremor severity | 72 weeks
  Change from pre to post-BoNT-A treatments in maximum angular tremor amplitude at the wrist in each treated arm. Angular tremor amplitude is one parameter reflecting the vectoral intensity of tremor segmented at each arm joint

SECONDARY OUTCOMES:
Clinical tremor severity | 72 weeks
  Improvement in upper limb tremor severity as determined by an increase >8 points on a standardized clinical assessment tool (Fahn-Tolosa-Marin Tremor Assessment Scale) pre and post Xeomin® injection using kinematic-determined injection parameters in both ET upper limbs
Accelerometric kinematic tremor severity | 72 weeks
  Change from pre and post-BoNT-A treatments in maximum log-transformed accelerometric tremor amplitude at wrist level (injected limb). Log-transformed accelerometric tremor amplitude is one parameter reflecting the non-vectoral intensity of tremor.
Quality of life measures | 72 weeks
  Quality of life for essential tremor questionnaire is used to measure the patient's impression of change due to treatment and its change on their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — LHSC
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Schantz EJ, Johnson EA. Properties and use of botulinum toxin and other microbial neurotoxins in medicine. Microbiol Rev. 1992 Mar;56(1):80-99. doi: 10.1128/mr.56.1.80-99.1992. PMID 1579114
- [Background] Evidente VG, Adler CH. An update on the neurologic applications of botulinum toxins. Curr Neurol Neurosci Rep. 2010 Sep;10(5):338-44. doi: 10.1007/s11910-010-0129-z. PMID 20567945
- [Background] Benito-Leon J, Louis ED. Essential tremor: emerging views of a common disorder. Nat Clin Pract Neurol. 2006 Dec;2(12):666-78; quiz 2p following 691. doi: 10.1038/ncpneuro0347. PMID 17117170
- [Background] Gironell A, Kulisevsky J. Diagnosis and management of essential tremor and dystonic tremor. Ther Adv Neurol Disord. 2009 Jul;2(4):215-22. doi: 10.1177/1756285609104791. PMID 21179530
- [Background] Jankovic J, Schwartz K, Clemence W, Aswad A, Mordaunt J. A randomized, double-blind, placebo-controlled study to evaluate botulinum toxin type A in essential hand tremor. Mov Disord. 1996 May;11(3):250-6. doi: 10.1002/mds.870110306. PMID 8723140
- [Background] Brin MF, Lyons KE, Doucette J, Adler CH, Caviness JN, Comella CL, Dubinsky RM, Friedman JH, Manyam BV, Matsumoto JY, Pullman SL, Rajput AH, Sethi KD, Tanner C, Koller WC. A randomized, double masked, controlled trial of botulinum toxin type A in essential hand tremor. Neurology. 2001 Jun 12;56(11):1523-8. doi: 10.1212/wnl.56.11.1523. PMID 11402109
- [Background] Adler CH, Bansberg SF, Hentz JG, Ramig LO, Buder EH, Witt K, Edwards BW, Krein-Jones K, Caviness JN. Botulinum toxin type A for treating voice tremor. Arch Neurol. 2004 Sep;61(9):1416-20. doi: 10.1001/archneur.61.9.1416. PMID 15364688
- [Background] Zesiewicz TA, Elble R, Louis ED, Hauser RA, Sullivan KL, Dewey RB Jr, Ondo WG, Gronseth GS, Weiner WJ; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter: therapies for essential tremor [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2005 Jun 28;64(12):2008-20. doi: 10.1212/01.WNL.0000163769.28552.CD. Epub 2005 Jun 22. PMID 15972843